CLINICAL TRIAL: NCT03181646
Title: Role of Citicoline in Treatment of Newborns With Hypoxic Ischemic Encephalopathy
Acronym: citicoline
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Fellow Neonatology Department, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITICOLINE
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): newborns with hypoxic ischemic encephalopathy grade 2/3 who will receive only supportive care
- study group (Experimental): newborns with hypoxic ischemic encephalopathy grade 2/3 who will receive citicoline along with supportive care
  Interventions: Drug: citicoline

INTERVENTIONS:
Drug: citicoline — intravenous citicoline 15 mg per kg per dose BD will be given to babies until oral feeds are established
  Arms: study group

SUMMARY:
Citicoline, is a naturally occurring compound and an intermediate in the metabolism of phosphatidylcholine. Phosphatidylcholine is an important component of the phospholipids of the cell membranes. Citicoline is composed of two molecules: cyti¬dine and choline. Both these molecules enter the brain separately and by passing through the blood-brain barrier where they act as substrates for intracellular synthesis of CDP-choline . This drug has been widely used in adults who suffer from acute ischemic strokes for than 4 decades with good results and has been proved to have a very good safety profile as well. It has various therapeutic effects at several stages of the ischemic cascade in acute ischemic stroke.

1. It stabilizes cell membranes by increasing phosphatidylcholine and sphingomyelin synthesis and by inhibiting the release of free fatty acids . By protecting membranes, citicoline inhibits glutamate release during ischemia. In an experimental model of ischemia in the rat, citicoline treatment decreased glutamate levels and stroke size.
2. Citicoline favors the synthesis of nucleic acids, proteins, acetylcholine and other neurotransmitters, and decreases free radical formation Therefore, citicoline simultaneously inhibits different steps of the ischemic cascade protecting the injured tissue against early and delayed mechanisms responsible for ischemic brain injury.
3. citicoline may facilitate recovery by enhancing synaptic outgrowth and increased neuroplasticity with decrease of neurologic deficits and improvement of behavioral performance.

Considering these pharmacologic properties of citicoline, we are planning to see its effects in newborns who have HIE which causes a global acute ischemic changes in developing brain.

ELIGIBILITY:
Inclusion Criteria:

* • Newborn babies having grade 2 and 3 HIE, of both genders delivered in labor room or operation theatre of our hospital.

  * Outdoor patients presenting within 24 hours of delivery

Exclusion Criteria:

* • Outborn babies presenting after 24 hours of delivery.

  * Patients with severe congenital malformations
  * Babies born extremely prematurely (less than 28 weeks)

Ages: 1 Hour to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2017-12-15 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
effect on sucking | 06 months after start of study
  time to establish full oral feeds
discharge time | 06 months after start of study
  time to discharge from hospital
effect on seizures | 06 months after start of study
  duration of seizures

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Rawalpindi, Punjab Province, Pakistan